CLINICAL TRIAL: NCT01782222
Title: A Multicenter, Multinational, Double-Blind, Placebo-Controlled, 3-Arm, Phase 4 Study To Evaluate The Efficacy Of Rotigotine On Parkinson's Disease-Associated Apathy, Motor Symptoms, And Mood
Brief Title: Trial to Evaluate The Efficacy Of Rotigotine on Parkinson's Disease-Associated Motor Symptoms And Apathy
Acronym: BRIGHT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PD0005; 2012-002840-26 (EudraCT Number)
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-07

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's Disease; Rotigotine; Apathy; Nonmotor; Motor; Neupro
MeSH Terms: conditions — Parkinson Disease; Lethargy | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rotigotine, high dose (Experimental): Rotigotine, transdermal patches, maximal 16 mg / 24 hours for patients with advanced Parkinson's Disease and 8 mg / 24 hours for those with early Parkinson's Disease
  Interventions: Drug: Rotigotine
- Rotigotine, low dose (Experimental): Rotigotine, transdermal patches, optimal dose, maximal 8 mg / 24 hours for patients with advanced Parkinson's Disease and 6 mg / 24 hours for those with early Parkinson's Disease
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator): Placebo transdermal patches
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rotigotine — Rotigotine, transdermal patches:
  10 cm^2 (2 mg / 24 hours); 20 cm^2 (4 mg / 24 hours); 30 cm^2 (6 mg / 24 hours); 40 cm^2 (8 mg / 24 hours)
  The maximum Rotigotine dose allowed is 8 mg / 24 hours or 16 mg / 24 hours for patients with advanced Parkinson's Disease and 6 mg / 24 hours or 8 mg / 24 hours for those with early Parkinson's Disease Duration: up to 21 weeks (including de-escalation)
  Other Names: (6S)-6-propyl-[2 (2 thienyl)ethyl]amino-5,6,7,8-tetrahydro-1-naphthalenol
  Arms: Rotigotine, high dose; Rotigotine, low dose
Other: Placebo — Placebo, matching transdermal patches
  Duration: up to 21 weeks (including de-escalation)
  Arms: Placebo

SUMMARY:
This trial is being conducted to assess the effects of Rotigotine over Placebo on improvement of Apathy and motor symptoms in subjects with early-stage and advanced stage idiopathic Parkinson´s Disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early or advanced idiopathic Parkinson's Disease
* Patients with advanced idiopathic Parkinson's Disease: intake of Levodopa on a stable dose of at least 200 mg/day
* Unsatisfactory control of Parkinson's Disease motor symptoms under current treatment
* Patients experiencing Apathy associated with Parkinson's Disease
* Hoehn and Yahr stage score of I to IV
* Mini-Mental State Examination score ≥ 25
* If an antidepressant drug is taken, the dose must be stable

Exclusion Criteria:

* Therapy with a Dopamine agonist
* Discontinuation from pervious therapy with a dopamine agonist after an adequate length of treatment, at adequate dose, due to lack of efficacy
* Any medical or psychiatric condition that jeopardizes / compromises patient's ability for participation
* Patient has received Neuroleptics, Dopamine releasing substances, Dopamine modulating substances, Alpha-Methyldopa, Metoclopramide, MAO-A inhibitors, Budipine, or Tolcapone
* Electroconvulsive therapy
* Patient has a

  * current/anticipated psychotherapy or behavior therapy
  * history of deep brain stimulation
  * history of suicide attempt or has suicidal ideation
  * impulse control disorder
  * severe Depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (42):
- United States (25):
  - 4320, Birmingham, Alabama
  - 4309, Oxnard, California
  - 4306, Ormond Beach, Florida
  - 4311, Palm Beach Gardens, Florida
  - 4313, Tampa, Florida
  - 4314, Decatur, Georgia
  - 4318, Chicago, Illinois
  - 4316, Winfield, Illinois
  - 4322, Des Moines, Iowa
  - 4304, Kansas City, Kansas
  - 4326, Springfield, Massachusetts
  - 4330, Ocean Springs, Mississippi
  - 4302, Las Vegas, Nevada
  - 4303, Commack, New York
  - 4317, New York, New York
  - 4323, New York, New York
  - 4319, Asheville, North Carolina
  - 4325, Charlotte, North Carolina
  - 4329, Akron, Ohio
  - 4312, Cincinnati, Ohio
  - 4324, Beaufort, South Carolina
  - 4332, Charleston, South Carolina
  - 4305, San Antonio, Texas
  - 4307, Salt Lake City, Utah
  - 4333, Virginia Beach, Virginia
- Austria (2):
  - 3001, Innsbruck
  - 3003, Linz
- Hungary (2):
  - 3301, Budapest
  - 3302, Debrecen
- Poland (3):
  - 3509, Gdansk
  - 3506, Gdynia
  - 3504, Poznan
- Slovakia (4):
  - 3801, Banská Bystrica
  - 3805, Bratislava
  - 3806, Krompachy
  - 3807, Žilina
- 3901, Ljubljana, Slovenia
- Spain (5):
  - 4001, Barcelona
  - 4006, Barcelona
  - 4009, Oviedo
  - 4005, Seville
  - 4010, Seville

REFERENCES:
- [Derived] Hauser RA, Slawek J, Barone P, Dohin E, Surmann E, Asgharnejad M, Bauer L. Evaluation of rotigotine transdermal patch for the treatment of apathy and motor symptoms in Parkinson's disease. BMC Neurol. 2016 Jun 7;16:90. doi: 10.1186/s12883-016-0610-7. PMID 27267880
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was planned to be conducted globally with 480 subjects (160 subjects per treatment group for the Full Analysis Set). Approx. 600 subjects were planned for enrollment in order to obtain 504 subjects for randomization. Subjects were randomized in a 1:1:1 ratio to either Rotigotine low dose, Rotigotine high dose or Placebo.
Pre-assignment Details: The Participant Flow refers to the Randomized Set (RS). The RS included all subjects who were randomized.
  The outcome of the Interim Analysis was to stop the study, i.e. no more subjects were enrolled into the study and all included subjects completed the study as planned.
Groups:
- Placebo: Placebo transdermal patches
  Placebo: Placebo, matching transdermal patches
  Duration: up to 21 weeks (including de-escalation)
- Rotigotine, Low Dose: Rotigotine, transdermal patches, optimal dose, maximal 8 mg / 24 hours for patients with advanced Parkinson's Disease and 6 mg / 24 hours for those with early Parkinson's Disease
  Rotigotine: Rotigotine, transdermal patches:
  10 cm^2 (2 mg / 24 hours); 20 cm^2 (4 mg / 24 hours); 30 cm^2 (6 mg / 24 hours); 40 cm^2 (8 mg / 24 hours)
  The maximum Rotigotine dose allowed was 8 mg / 24 hours for patients with advanced Parkinson's Disease and 6 mg / 24 hours for those with early Parkinson's Disease Duration: up to 21 weeks (including de-escalation)
- Rotigotine, High Dose: Rotigotine, transdermal patches, maximal 16 mg / 24 hours for patients with advanced Parkinson's Disease and 8 mg / 24 hours for those with early Parkinson's Disease
  Rotigotine: Rotigotine, transdermal patches:
  10 cm^2 (2 mg / 24 hours); 20 cm^2 (4 mg / 24 hours); 30 cm^2 (6 mg / 24 hours); 40 cm^2 (8 mg / 24 hours)
  The maximum Rotigotine dose allowed was 16 mg / 24 hours for patients with advanced Parkinson's Disease and 8 mg / 24 hours for those with early Parkinson's Disease Duration: up to 21 weeks (including de-escalation)
Period: Overall Study
Arm/Group | Placebo | Rotigotine, Low Dose | Rotigotine, High Dose
Started | 40 | 41 | 41
Completed | 32 | 30 | 37
Not Completed | 8 | 11 | 4
Not completed — Adverse Event | 4 | 5 | 3
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 1
Not completed — Moved to other state | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population refers to the Safety Set (SS). The SS included all randomized subjects who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rotigotine, Low Dose | Rotigotine, High Dose | Total
Number analyzed (Participants) | 40 | 41 | 41 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (11.7) | 68.1 (10.5) | 70.2 (8.0) | 69.1 (10.1)
Age, Customized [Number; unit: participants]
  >18 - < 65 years | 14 | 17 | 12 | 43
  ≥ 65 years | 26 | 24 | 29 | 79
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 14 | 46
  Male | 22 | 27 | 27 | 76
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 1 | 2 | 1 | 4
  White | 38 | 39 | 40 | 117
  Other/mixed | 1 | 0 | 0 | 1
Weight [Mean (Standard Deviation); unit: kilograms] | 79.59 (14.73) | 77.34 (17.93) | 78.96 (15.96) | 78.62 (16.17)
Height [Mean (Standard Deviation); unit: centimeters] | 167.16 (10.34) | 169.25 (10.76) | 170.88 (10.94) | 169.10 (10.70)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter] | 28.53 (4.79) | 26.86 (4.89) | 26.90 (3.86) | 27.42 (4.57)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End of the Maintenance Period in the Score of the Apathy Evaluation Scale (AS) Rated by the Patient
Description: The Apathy Scale (AS) is an abbreviated version of the Apathy Evaluation Scale. The AS (Starkstein et al, 1992) consists of 14 items phrased as questions by the examiner that are to be answered on a 4-point Likert scale. It was developed specifically for subjects with Parkinson's disease because the Apathy Evaluation Scale was considered too demanding.
  The questions comprising the AS were answered by the subject. The total scores for Apathy Evaluation Scale ranges from 0 (best possible outcome) to 42 (worst possible outcome).
Time Frame: Baseline (Visit 2) until End of the Maintenance Period / Early Withdrawal (up to 19 weeks after Baseline)
Population: The Analysis Population refers to the Full Analysis Set (FAS). The FAS included all subjects who were randomized, received at least 1 dose of study medication, and had a valid primary efficacy Baseline measurement and at least 1 valid post-Baseline Maintenance or valid Withdrawal primary efficacy measurement for both primary efficacy variables.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine, Low Dose | Rotigotine, High Dose
Number analyzed (Participants) | 40 | 36 | 40
scores on a scale | -4.4 (4.9) | -4.6 (6.7) | -4.9 (5.9)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine, Low Dose; Test type: Superiority or Other; p = 0.977, ANCOVA; ANCOVA model for the change from Baseline to End of Maintenance containing treatment and disease stage as factors, and Baseline value as covariate; Least Square Mean = 0.04, 95% CI 2-sided [-2.42 to 2.50], Standard Error of Mean 1.24
Statistical Analysis 2: Comparison: Placebo vs Rotigotine, High Dose; Test type: Superiority or Other; p = 0.859, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -0.22, 95% CI 2-sided [-2.61 to 2.18], Standard Error of Mean 1.21

2. Primary Outcome: Change From Baseline to the End of the Maintenance Period in the Total Score of the Unified Parkinson's Disease Rating Scale (UPDRS) Parts II (Activities of Daily Living) + III (Motor Symptoms)
Description: Part II of the Unified Parkinson's Disease Rating Scale (UPDRS) assesses the subject's activities of daily living. Part III assesses motor function. The UPDRS is completed by questioning the subject about his/her general state in conjunction with any observations made by the investigator (or designee) since the previous visit. Part II is subject-rated and Part III is physician-rated. The UPDRS Part II (Activities of Daily Living) consists of 13 items scored between 0 and 4. The sum score was calculated as the sum of these 13 individual scores. The UPDRS Part III (motor subscale) consists of 27 items and sub items scored between 0 and 4. The sum score was calculated as sum of these 27 individual scores. The sum score of UPDRS Parts II and III is the sum of the corresponding single sum scores. A negative value indicates an improvement.
Time Frame: Baseline (Visit 2) until End of the Maintenance Period / Early Withdrawal (up to 19 weeks after Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine, Low Dose | Rotigotine, High Dose
Number analyzed (Participants) | 40 | 36 | 40
scores on a scale | -4.8 (10.4) | -12.4 (14.0) | -10.7 (8.4)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine, Low Dose; Test type: Superiority or Other; p = 0.005, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -7.29, 95% CI 2-sided [-12.30 to -2.28], Standard Error of Mean 2.53
Statistical Analysis 2: Comparison: Placebo vs Rotigotine, High Dose; Test type: Superiority or Other; p = 0.015, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -6.06, 95% CI 2-sided [-10.90 to -1.21], Standard Error of Mean 2.45

3. Secondary Outcome: Change From Baseline to the End of the Maintenance Period in the Score of the Apathy Evaluation Scale (AS) Rated by the Caregiver (Where Available)
Description: The Apathy Scale (AS) is an abbreviated version of the Apathy Evaluation Scale. The AS (Starkstein et al, 1992) consists of 14 items phrased as questions by the examiner that are to be answered on a 4-point Likert scale. It was developed specifically for subjects with Parkinson's disease because the Apathy Evaluation Scale was considered too demanding.
  The questions comprising the AS were answered by the caregiver. The questions were asked in a structured interview format. The caregiver was interviewed by appropriate medical staff and asked questions about the subject in the third person.The total scores for Apathy Evaluation Scale ranges from 0 (best possible outcome) to 42 (worst possible outcome).
Time Frame: Baseline (Visit 2) until End of the Maintenance Period / Early Withdrawal (up to 19 weeks after Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine, Low Dose | Rotigotine, High Dose
Number analyzed (Participants) | 16 | 16 | 13
scores on a scale | -1.5 (7.0) | -4.8 (8.0) | -5.5 (6.1)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine, Low Dose; Test type: Superiority or Other; p = 0.200, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -3.20, 95% CI 2-sided [-8.17 to 1.76], Standard Error of Mean 2.46
Statistical Analysis 2: Comparison: Placebo vs Rotigotine, High Dose; Test type: Superiority or Other; p = 0.239, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -3.04, 95% CI 2-sided [-8.19 to 2.10], Standard Error of Mean 2.55

4. Secondary Outcome: Change From Baseline to the End of the Maintenance Period in the Sum Score of the 8-item Parkinson's Disease Questionnaire (PDQ-8)
Description: The 8-Item Parkinson's Disease Questionnaire (PDQ-8) (Peto et al, 1998) is a self-administered questionnaire that provides a reliable measure of overall health status. The PDQ-8 collects 8 items with 5 categories each (0=never, 1=occasionally, 2=sometimes, 3=often, 4=always or cannot do at all). The total score was calculated by summing the scores of all applicable questions and convert the resulting sum to a summary index score between 0 and 100 by multiplying with 100/32. A negative value indicates an improvement.
Time Frame: Baseline (Visit 2) until End of the Maintenance Period / Early Withdrawal (up to 19 weeks after Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine, Low Dose | Rotigotine, High Dose
Number analyzed (Participants) | 40 | 36 | 40
scores on a scale | -3.8 (14.0) | -5.1 (20.4) | -10.0 (15.0)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine, Low Dose; Test type: Superiority or Other; p = 0.519, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -2.09, 95% CI 2-sided [-8.48 to 4.31], Standard Error of Mean 3.23
Statistical Analysis 2: Comparison: Placebo vs Rotigotine, High Dose; Test type: Superiority or Other; p = 0.111, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -5.06, 95% CI 2-sided [-11.29 to 1.17], Standard Error of Mean 3.15

5. Secondary Outcome: Change From Baseline to the End of the Maintenance Period in the Sum Score of the Mood / Cognition Domain of the Nonmotor Symptom Assessment Scale (NMSS)
Description: Nonmotor performance was assessed via the Nonmotor Symptom Assessment Scale (NMSS), an accepted scale that has been validated in an international study (Naidu et al, 2006; Chaudhuri et al, 2007), at the Baseline Visit as well as at the end of the Maintenance Period. The severity and frequency of the subject's nonmotor symptoms were assessed by the investigator (or designee) in the following 9 domain categories: cardiovascular, including falls; sleep/fatigue; mood/cognition; perceptual problems/hallucinations; attention/memory; gastrointestinal tract; urinary; sexual function; and miscellaneous.
  Items are scored for severity (from 0 (none) to 3 (severe)) and frequency (from 1 (rarely) to 4 (very frequent )). The score was calculated as severity x frequency. The theoretical minimum is 0 (best possible outcome) and maximum total score is 360 points (worst possible outcome).
Time Frame: Baseline (Visit 2) until End of the Maintenance Period / Early Withdrawal (up to 19 weeks after Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine, Low Dose | Rotigotine, High Dose
Number analyzed (Participants) | 39 | 32 | 39
scores on a scale | -4.6 (7.9) | -9.8 (12.1) | -9.8 (10.7)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine, Low Dose; Test type: Superiority or Other; p = 0.060, ANCOVA; ANCOVA model for the change from Baseline to End of Treatment containing treatment and disease stage as factors, and Baseline value as covariate; Least Square Mean = -3.62, 95% CI 2-sided [-7.39 to 0.15], Standard Error of Mean 1.90
Statistical Analysis 2: Comparison: Placebo vs Rotigotine, High Dose; Test type: Superiority or Other; p = 0.034, ANCOVA; [statistical method as in outcome 5, analysis 1]; Least Square Mean = -3.88, 95% CI 2-sided [-7.46 to -0.30], Standard Error of Mean 1.80

6. Secondary Outcome: Change From Baseline to the End of the Maintenance Period in the Sum Score of the Snaith Hamilton Pleasure Scale (SHAPS)
Description: The Snaith Hamilton Pleasure Scale (SHAPS) (Snaith et al, 1995) is a self-report instrument developed for the assessment of hedonic capacity. The sum of the 14 items scores range from 0 to 14. A higher score represents more anhedonic symptoms.
Time Frame: Baseline (Visit 2) until End of the Maintenance Period / Early Withdrawal (up to 19 weeks after Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine, Low Dose | Rotigotine, High Dose
Number analyzed (Participants) | 40 | 36 | 40
scores on a scale | -0.5 (2.5) | -1.3 (2.2) | -0.9 (2.8)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine, Low Dose; Test type: Superiority or Other; p = 0.334, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -0.38, 95% CI 2-sided [-1.16 to 0.40], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Placebo vs Rotigotine, High Dose; Test type: Superiority or Other; p = 0.968, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = 0.02, 95% CI 2-sided [-0.74 to 0.77], Standard Error of Mean 0.38

7. Secondary Outcome: Change From Baseline to the End of the Maintenance Period in the Sum Score of the Beck Depression Inventory Second Edition (BDI-II)
Description: The Beck Depression Inventory (BDI) is a self-report instrument to measure depression symptoms and severity (Beck et al, 1961). The BDI-II is a revised version of the scale in order to be more consistent with the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for depression (Beck et al, 1996). There are 21 items in the BDI-II, classified as cognitive-affective (Items 1-13) and somatic-performance (Items 14-21) subscales. The degree of severity is indicated on a 4-point scale; items are rated from 0 (not at all) to 3 (extreme form of each symptom). Scores of 0-13 indicate minimal depression, 14-19 indicate mild depression, 20-28 indicate moderate depression, and 29-63 indicate severe depression.
Time Frame: Baseline (Visit 2) until End of the Maintenance Period / Early Withdrawal (up to 19 weeks after Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine, Low Dose | Rotigotine, High Dose
Number analyzed (Participants) | 39 | 31 | 39
scores on a scale | -3.3 (7.0) | -2.9 (5.9) | -3.7 (5.3)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine, Low Dose; Test type: Superiority or Other; p = 0.899, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = 0.16, 95% CI 2-sided [-2.34 to 2.66], Standard Error of Mean 1.26
Statistical Analysis 2: Comparison: Placebo vs Rotigotine, High Dose; Test type: Superiority or Other; p = 0.785, ANCOVA; [statistical method as in outcome 5, analysis 1]; Least Square Mean = -0.33, 95% CI 2-sided [-2.68 to 2.03], Standard Error of Mean 1.19

8. Secondary Outcome: Change From Baseline to the End of the Maintenance Period in the Sum Score of the Unified Parkinson's Disease Rating Scale (UPDRS) Part III (Motor Subscale) in "on" State
Description: Part III of the Unified Parkinson's Disease Rating Scale (UPDRS) assesses motor function. The UPDRS is completed by questioning the subject about his/her general state in conjunction with any observations made by the investigator (or designee) since the previous visit.
  The UPDRS Part III (motor subscale) had to be measured in the "on" state and consisted of 27 items and sub items scored between 0 and 4. The sum score ranged between 0 and 108 and was calculated as sum of the 27 individual scores. If 1 or more items were missing and could not be substituted with a previous post-Baseline value, the sum score was also missing.
  A negative value indicates an improvement.
Time Frame: Baseline (Visit 2) until End of the Maintenance Period / Early Withdrawal (up to 19 weeks after Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine, Low Dose | Rotigotine, High Dose
Number analyzed (Participants) | 40 | 36 | 40
scores on a scale | -3.4 (8.2) | -8.9 (10.4) | -8.1 (7.3)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine, Low Dose; Test type: Superiority or Other; p = 0.014, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -4.96, 95% CI 2-sided [-8.91 to -1.01], Standard Error of Mean 1.99
Statistical Analysis 2: Comparison: Placebo vs Rotigotine, High Dose; Test type: Superiority or Other; p = 0.013, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -4.83, 95% CI 2-sided [-8.63 to -1.03], Standard Error of Mean 1.92

9. Secondary Outcome: Change From Baseline to the End of the Maintenance Period in the Score of the Clinical Global Impression Scale (CGI) Item I (Severity of Illness)
Description: The Clinical Global Impression (CGI) scales (Guy and Bonato, 1970) were initially developed for a risk-benefit estimation within the treatment of mentally ill patients. The 4 global scales (severity of illness, change in severity from Baseline, therapeutic efficacy, and tolerability of treatment) are used as different measures of treatment outcome in different kinds of pharmacological studies.
  The CGI Item 1 (severity of illness) collected 1 answer out of 8 categories (0-'Not assessed', 1-'Normal, not at all ill', 2-'Borderline ill', 3-'Mildly ill', 4-'Moderately ill', 5-'Markedly ill', 6-'Severely ill', and 7-'Among the most extremely ill patients') at each assessment. The category 0-'Not assessed' was considered as missing and therefore used neither for calculation nor for display purposes.
Time Frame: Baseline (Visit 2) until End of the Maintenance Period/Early Withdrawal (up to 19 weeks after Baseline)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Rotigotine, Low Dose | Rotigotine, High Dose
Number analyzed (Participants) | 40 | 36 | 40
participants
  Normal, not ill at all | 1 | 1 | 2
  Borderline ill | 6 | 2 | 3
  Mildly ill | 19 | 16 | 21
  Moderately ill | 9 | 10 | 12
  Markedly ill | 2 | 1 | 1
  Severely ill | 1 | 1 | 0
  Amongst the most extremely ill subjects | 0 | 0 | 0
  Missing | 2 | 5 | 1

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAEs) were reported from Baseline up to the Safety Follow-up Visit (approximately during 19 weeks).
Description: The Baseline Analysis Population refers to the Safety Set (SS). The SS includes all randomized subjects who received at least 1 dose of study medication.
Groups:
- Rotigotine, Low Dose: Rotigotine, transdermal patches, optimal dose, maximal 8 mg / 24 hours for patients with advanced Parkinson's Disease and 6 mg / 24 hours for those with early Parkinson's Disease
  Rotigotine: Rotigotine, transdermal patches:
  10 cm^2 (2 mg / 24 hours); 20 cm^2 (4 mg / 24 hours); 30 cm^2 (6 mg / 24 hours); 40 cm^2 (8 mg / 24 hours)
  Optimal dosage:
  The maximum Rotigotine dose allowed was 8 mg / 24 hours or 16 mg / 24 hours for patients with advanced Parkinson's Disease and 6 mg / 24 hours or 8 mg / 24 hours for those with early Parkinson's Disease Duration: up to 21 weeks (including de-escalation)
- Rotigotine, High Dose: Rotigotine, transdermal patches, maximal 16 mg / 24 hours for patients with advanced Parkinson's Disease and 8 mg / 24 hours for those with early Parkinson's Disease
  Rotigotine: Rotigotine, transdermal patches:
  10 cm^2 (2 mg / 24 hours); 20 cm^2 (4 mg / 24 hours); 30 cm^2 (6 mg / 24 hours); 40 cm^2 (8 mg / 24 hours)
  Optimal dosage:
  The maximum Rotigotine dose allowed was 8 mg / 24 hours or 16 mg / 24 hours for patients with advanced Parkinson's Disease and 6 mg / 24 hours or 8 mg / 24 hours for those with early Parkinson's Disease Duration: up to 21 weeks (including de-escalation)
Arm/Group | Placebo | Rotigotine, Low Dose | Rotigotine, High Dose
Serious Adverse Events (participants affected / at risk) | 4/40 | 2/41 | 1/41
Other Adverse Events (participants affected / at risk) | 18/40 | 17/41 | 15/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Rotigotine, Low Dose (N=41) | Rotigotine, High Dose (N=41)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Rotigotine, Low Dose (N=41) | Rotigotine, High Dose (N=41)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (5) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Application site pruritus (General disorders) | 2 (2) | 4 (4) | 1 (2)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 3 (3) | 2 (2)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2) | 4 (5)
Dyskinesia (Nervous system disorders) | 2 (3) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 4 (6) | 1 (1) | 3 (6)
Depression (Psychiatric disorders) | 2 (2) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6) | 1 (1) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days